CLINICAL TRIAL: NCT01579487
Title: Non-Invasive Reduction of Abdominal Fat Utilizing the JUNO Applicator
Brief Title: Extended Follow-Up Study for Subjects Who Participated in 2010 Study
Acronym: JUNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA10-001.A1-EXT
Record Dates: First submitted 2012-03-15; First posted 2012-04-18 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2012-03

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Zeltiq System — This is a follow-up study from the initial treatments performed in 2010. No additional treatments will be performed.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
This study is being performed to follow up on subjects who participated in the initial study (ZA10-001) in 2010.

DETAILED DESCRIPTION:
The primary objective of this investigation is to assess the durability of treatment outcomes with the ZELTIQ System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject participated in the ZA10-001 study, and received all study treatments.
2. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Subject has had any surgical or aesthetic procedure(s) in or around the abdomen since the completion of the ZA10-001 study treatments.
2. Subject is pregnant.
3. Subject is unable or unwilling to comply with the study requirements.
4. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
5. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the integrity of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Independent Photo Review | 12+ mos post treatment
  The primary effectiveness endpoint is the correct identification of the series of pre-treatment images by the three reviewers.

SECONDARY OUTCOMES:
Access reduction | 12+ mos post treatment
  Reduction in the fat layer thickness
Subject Satisfaction | 12+ mos post treatment
  Subject satisfaction with the Zeltiq procedure as determined by the results of a subjects satisfaction questionnaire at the follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Flor Mayoral, MD, Principal Investigator — Mayoral Dermatology
Locations (1):
- Mayoral Dermatology, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No